CLINICAL TRIAL: NCT05426759
Title: Atrial Deganglionation as a Therapy for Cardiac Surgery Patients With Atrial Fibrillation
Acronym: Neural-AF-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrian Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-002
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GP Ablation (Experimental): Single arm study with GP ablations performed during open-chest surgery
  Interventions: Device: Pulsed Field Ablation of epicardial Ganglionated Plexi.

INTERVENTIONS:
Device: Pulsed Field Ablation of epicardial Ganglionated Plexi. — Using Pulsed Field Ablation (PFA), delivered via an epicardial catheter, to selectively ablate the ganglionated plexi (GP) on the epicardial surface of the heart.

SUMMARY:
A prospective single-arm study of ganglionated plexi ablation in cardiothoracic surgery patients with a history of atrial fibrillation.

DETAILED DESCRIPTION:
This study assesses the use of electroporation/pulsed field ablation (PFA) to selectively ablate ganglionated plexi in cardiothoracic surgery patients with atrial fibrillation. The PFA treatment will be performed in up to 12 patients with a history of paroxysmal atrial fibrillation. The primary end point will be recurrence of atrial fibrillation out to 1 year follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 70 years.
* Scheduled for open-chest cardiothoracic surgery, for coronary artery bypass grafting and/or aortic valve repair/replacement
* Have a documented medical history of paroxysmal or early-stage persistent atrial fibrillation within the previous 12 months.
* Legally competent and willing to sign the informed consent.
* Life expectancy of at least 2 years.

Exclusion Criteria:

* Previous cardiac surgery
* Prior pericardial interventions
* Prior endocardial or epicardial pulmonary vein isolation (PVI), or any other invasive AF therapy
* Previous or existing pericarditis
* Use of amiodarone within the previous 12 months.
* Long-standing persistent atrial fibrillation
* Indication for mitral or tricuspid valve surgery
* Indication for concomitant left atrial appendage (LAA) ligation or excision
* History of previous radiation therapy on the thorax
* History of previous thoracotomy.
* Prior electrical or mechanical isolation of the Left Atrial Appendage (LAA)
* The presence of LAA occlusion devices, coronary stents, prosthetic heart valves, pacemakers or implantable cardioverter defibrillators (ICDs)
* Myocardial infarction within the previous 2 months
* New York Heart Association (NYHA) Class IV heart failure symptoms
* Left Ventricular Ejection Fraction (LVEF) < 40%, measured by transthoracic echocardiography (TTE)
* Left atrial diameter > 5.0 cm, measured by transthoracic echocardiography (TTE)
* The presence of left atrial thrombus when examined by transesophageal echocardiography (TEE)
* The presence of atrial fibrillation (AF) attributable to non-cardiovascular causes such as thyroid disease, electrolyte imbalance/dehydration or other reversible causes
* Active infection or sepsis as evidenced by increased white blood cell count, elevated C-reactive protein (CRP) or temperature > 38.5°C
* Known or documented carotid stenosis > 80%
* Stroke or transient ischemic attack within the previous 6 months
* Known or documented epilepsy
* Pregnancy or child-bearing potential without adequate contraception
* Circumstances that prevent follow-ups
* Drug abuse
* Patients cannot be enrolled in another clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tbilisi Heart & Vascular Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ganglionated Plexi Ablation: Single arm study with Ganglionated Plexi (GP) ablations performed during open-chest cardiothoracic surgery. Ablation is performed using pulsed electric fields, delivered via an epicardial catheter, to selectively ablate the GPs on the epicardial surface of the heart.
Period: Overall Study
Arm/Group | Ganglionated Plexi Ablation
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ganglionated Plexi Ablation
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Left Atrial Diameter [Mean (Standard Deviation); unit: cm] | 3.6 (0.6)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: % (of total left ventricle volume)] | 48.4 (4.4)
Hypertension [Count of Participants; unit: Participants] | 12
Diabetes [Count of Participants; unit: Participants] | 0
Stroke or Transient Ischemic Attack [Count of Participants; unit: Participants] | 0
Myocardial Infarction [Count of Participants; unit: Participants] | 3
Paroxysmal Atrial Fibrillation [Count of Participants; unit: Participants] | 12
Valve Disease [Count of Participants; unit: Participants] | 2
Beta Blockers [Count of Participants; unit: Participants] | 12
Anti-Arrhythmic Drugs [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients in Sinus Rhythm at 12 Months.
Description: Patients will be monitored with 24 hour Holter at 12 months
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Ganglionated Plexi Ablation
Number analyzed (Participants) | 12
Participants | 12

2. Secondary Outcome: Extension of AERP
Description: The acute increase in atrial effective refractory period (AERP) i.e. by comparing AERP values from immediately before and immediately after ablation.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Ganglionated Plexi Ablation
Number analyzed (Participants) | 10
ms | 12 (41)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ganglionated Plexi Ablation
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganglionated Plexi Ablation (N=12)
Atrial bleed (Cardiac disorders) | 1 — During ablation at the ligament of Marshall, a left atrial effusion was noted by the surgeon. This was immediately sutured and no further issues were noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT05426759/Prot_SAP_000.pdf